CLINICAL TRIAL: NCT05679180
Title: Navigated Microsecond Laser for Chronic Central Serous Chorioretinopathy: MICROPULSE
Acronym: MICROPULSE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study withdrawn by clinical team
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2021/39
Record Dates: First submitted 2022-12-28; First posted 2023-01-10 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Central Serous Chorioretinopathy
Keywords: retina; photodynamic therapy; micropulse laser; central serous chorioretinopathy
MeSH Terms: conditions — Central Serous Chorioretinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- micropulse laser (Experimental): treatment with confluent spots over the area of focal leak on the earliest phase of fundus fluorescein angiography on Navilas® system using 5% duty cycle with 100 micron spot size with 200 ms envelope. Thirty percent of threshold laser burn power was used.
  Interventions: Device: micropulse laser

INTERVENTIONS:
Device: micropulse laser — treatment with confluent spots over the area of focal leak on the earliest phase of fundus fluorescein angiography on Navilas® system using 5% duty cycle with 100 micron spot size with 200 ms envelope. Thirty percent of threshold laser burn power was used.

SUMMARY:
MICROPULSE study aims to evaluate the efficacy of navigated microsecond laser (nMSL) for chronic central serous chorioretinopathy (CSCR).

DETAILED DESCRIPTION:
Chronic central serous chorioretinopathy (CSCR) is characterized by persistent subretinal fluid (SRF) and extensive outer retinal damage on optical coherence tomography (OCT). In the last years several treatment modalities for chronic CSCR have been investigated. These treatments have included pharmacologic therapy, photodynamic therapy (PDT) and microsecond laser.

PDT is the main treatment for CSCR, especially for chronic CSCR. But the efficacy of PDT is variable and could be associated with various complications such as retinal pigment epithelium (RPE) atrophy. Furthermore other limitations of PDT are unavailability and high cost.

Recently some studies have suggested an efficacy of micropulse laser in chronic CSCR, with stabilization of visual acuity, improvement in retinal sensitivity and without any complications.

The present study aims to evaluate the efficacy of a treatment by guided micropulse laser in the management of chronic CSCR. The efficacity will be evaluated 6 weeks and 3 months after the treatment on anatomical outcomes (central macular thickness in microns)

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* vision complaints for more than 6 weeks
* subretinal fluid confirmed on OCT
* diagnosis of CSCR confirmed by fluorescein and indocyanine green angiography
* Signed informed consent
* Affiliated or beneficiary of health insurance

Exclusion Criteria:

* History of treatment of CSC with other modalities (PDT, eplerenone) in the past 3 months
* Other macular conditions : Age-related Macular Degeneration (AMD), polypoidal vasculopathy, choroidal neovascularization
* Cataract or opacities interfering with acquisition or treatment
* Myopia> 6 diopter
* Visual acuity<20/200
* Treatment with steroids (per-os, inhaled or cutaneous) in the past 3 months
* Intra-vitreal injections of anti-VEGF (Vascular Endothelial Growth Factor) or steroids in the past 3 months
* History of allergy to fluorescein or indocyanine
* Inability to agree to participate to the study
* Pregnant or breastfeeding woman
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-11 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
central macular thickness | Month 3
  central macular thickness measured in microns and determined on spectral-domain OCT

SECONDARY OUTCOMES:
central retinal thickness | Baseline, Month 3
  central retinal thickness (micrometers)
visual acuity | Baseline, Month 3
  visual acuity via ETDRS (Early Treatment of Diabetic Retinopathy Study) scale. The EDTRS scale is expressed in number of letters read. The scale is logarithmic, i.e. the progression between the 14 lines is geometric (by a factor equal to the cube root of 2). A loss of 3 lines of visual acuity thus corresponds to a doubling of the visual angle.This allows to determine the necessary corrections (sphere, cylinder, axis
eye sensitivity | Baseline, Month 3
  eye sensitivity measured with microperimetry in decibels (dB)
presence of sub-retinal fluid | Baseline, Month 3
  presence of sub-retinal fluid on Spectral-Domain Optical Coherence Tomography (SD-OCT)
presence of intraretinal cysts | Baseline, Month 3
  presence of intraretinal cysts on SD-OCT
presence of flat irregular pigment epithelium detachment | Baseline, Month 3
  presence of flat irregular pigment epithelium detachment (FIPED) on SD-OCT
presence of neovascularization | Baseline, Month 3
  presence of type 1 neovascularization on OCT-angiography

IPD SHARING:
Plan to Share IPD: No